CLINICAL TRIAL: NCT03653611
Title: The CAPTURE Study: Validating a Unique Chronic Obstructive Pulmonary Disease (COPD) Case Finding Tool in Primary Care
Brief Title: The CAPTURE Study: Validating a Unique COPD Case Finding Tool in Primary Care (Aim 2)
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Michigan (Other); National Jewish Health (Other); Wake Forest University Health Sciences (Other); Duke University (Other); High Plains Research Network (Network); L.A. Net Community Health Resource Network (Other); Oregon Health and Science University (Other); University of Minnesota (Other); University of Kentucky (Other); COPD Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1803019032-2; R01HL136682-01 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-08-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; CAPTURE; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinician Participants: Two Aim 2 practices are selected by each of their 5 affiliated PBRNs based upon willingness to participate and variability of primary care practice type within the PBRN. Differences in practice size, staffing, ownership, prior quality improvement engagement, geography, patient population socioeconomic status (SES) or languages spoken are among the among the selection criteria the PBRNs will utilize to choose.
  Interventions: Other: On-site Practice Assessment; Other: Clinical Staff Questionnaires; Other: Modular online COPD Education; Other: COPD in Primary Care/CAPTURE Introduction Focus Groups
- Patient Participants: 200 patients, who are enrolled in Aim 1 (approximately 40 from each PBRN) will be invited to take a CAPTURE opinion survey
  Interventions: Other: Patient Opinion Surveys

INTERVENTIONS:
Other: On-site Practice Assessment — The assessment takes place in three parts; the pre-observation practice overview (conducted with the 2 practice clinicians - 60 minutes), the ½ day practice workflow observation (observation by one member of the Aim 2 research team of common and testing areas used for the respiratory patient). There is no patient engagement and no collection of patient-specific identification or health information), and the post-observation practice summary (conducted with the same 2 practice clinicians - 30 minutes).
  Groups: Clinician Participants
Other: Clinical Staff Questionnaires — Written or on-line questionnaires are provided to participating and consented staff personnel at two practice levels -- Non-Prescribing clinical (also known as "support") staff and Prescribing (PR) clinical (also known as "provider") staff.
  Groups: Clinician Participants
Other: Patient Opinion Surveys — 200 Eligible participants will complete a one-time 5 to 10 minute CAPTURE opinion survey.
  Groups: Patient Participants
Other: Modular online COPD Education — Access to free, COPD on-line, continuing education is provided for all clinical staff at each practice. Each module will take 20 minutes or less. Aim 2 clinician participant access and completion of COPD education modules is assessed by clinician questionnaires and focus group item response over 12 months (between months 2 and 14 of Aim 2 timeline).
  Groups: Clinician Participants
Other: COPD in Primary Care/CAPTURE Introduction Focus Groups — Two 45 to 60-minute focus group discussions occur at each Aim 2 practice. Focus groups are informed by practice demographics, practice assessment data, as well as patient opinion from CAPTURE surveys and past CAPTURE study. Focus group candidate themes and prompts are developed for non-prescribing clinical staff (NPR) and prescribing clinical staff (PR) and are presented at separate on-site focus group sessions to allow more detailed discussion of role responsibility in the context of daily practice workflow.
  Groups: Clinician Participants

SUMMARY:
This is a qualitative research exploration engaging clinical staff at all levels from 10 Practice-Based Research Networks (PBRNs) serving US patient populations of differing gender, racial, ethnic, urban/rural and socio-economic blends, in the incorporation of a one-page, five-item questionnaire with selective PEF measurement (CAPTURE).

DETAILED DESCRIPTION:
This is a prospective, multi-center qualitative study engaging clinical staff at all levels from primary care practices serving US patient populations of differing gender, racial, ethnic, urban/rural and socio-economic blends.

The CAPTURE tool consists of a 5-item self-administered questionnaire and selected use of peak expiratory flow (PEF) measurement, designed to identify clinically significant COPD.

This study will assess, using the RE-AIM approach, how real-word primary care practices might potentially use CAPTURE to: a) identify target populations (Reach); b) appraise optimal targeted respiratory history and symptoms consistent with clinically significant COPD (Effectiveness); c) integrate into practice workflow (Adoption); d) deliver changes and improvements to COPD care within the scope of real-world clinical practice (Implementation); and e) persist in use and quality over time (Maintenance).

Approximately 150 clinicians from 10 participating primary care practices will undergo detailed implementation investigation of the CAPTURE case finding model for clinically significant COPD. In addition, 200 enrolled participants will complete a 10-minute written CAPTURE opinion survey.

Using the RE-AIM framework and consistent phased qualitative analyses, this aim ascertains reach, impact, adoption, implementation and maintenance primary care feasibility recommendation characteristics of CAPTURE via pooled assessment of prescriber clinical staff, non-prescriber clinical staff, CAPTURE-eligible patients and local PBRN clinical quality improvement expertise from 10 primary care practices across 5 US regions.

ELIGIBILITY:
Inclusion Criteria:

Clinician Participants:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with availability and all study procedures for the duration of the study by the 10 practices (through PBRN recruitment) and their up to 15 clinicians within (through informed consent).
3. Male or female, aged 45 - 80 years

Patient participants [200 participants enrolled in Aim 1 of the CAPTURE Study for an opinion survey]:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 45 - 80 years.

Exclusion Criteria:

1. Clinician participants: current employment at practices participating in aims 1 and/or 3
2. Clinician participants: from practices providing fewer than 2 clinician participants
3. Patient participants: meeting the exclusion criteria for aims 1 and 3 (above)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practices participating in Aim 2, will be selected by each of their 5 affiliated PBRNs based upon willingness to participate and variability of primary care practice type within the PBRN. Differences in practice size, staffing, ownership, prior quality improvement engagement, geography, patient population socioeconomic status (SES) or languages spoken are among the among the selection criteria the PBRNs will utilize to choose.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Primary care clinician perspective on implementing CAPTURE into primary care practice. | Baseline to 2 years
  Primary care clinician perspective on implementing CAPTURE will be assessed using the RE-AIM approach in two focus group sessions consisting of clinical staff self-reporting current clinical practices, the process for implementing a new tool into practice and review of the CAPTURE tool.

SECONDARY OUTCOMES:
Primary care clinician knowledge about respiratory care at the provider level. | Baseline to 2 years
  Primary care clinician knowledge will be assessed using a questionnaire to self report about knowledge and beliefs regard Chronic Obstructive Pulmonary Disease (COPD) and COPD management.
Primary care clinician knowledge about respiratory care at the provider level. | Baseline to 2 years
  Primary care clinician knowledge will be assessed using two focus groups to self report on the staff's knowledge regarding respiratory care.
Primary care clinician attitudes and beliefs regarding respiratory care and communication within their current practice. | Baseline to 2 years
  Primary care clinician attitudes and beliefs will be assessed using a questionnaire to self report respiratory care in their current practice.
Primary care clinician self-efficacy in provider-specific respiratory clinical care. | Baseline to 2 years
  Primary care clinician self-efficacy will be assessed using two focus groups to self report on the staff's perspective regarding self-efficacy of provider-specific respiratory practices.
Primary care clinician attitudes and beliefs about clinical quality improvement and communication within their current practice. | Baseline to 2 years
  Primary care clinician attitudes and beliefs regarding quality improvement and communication within their current practice will be assessed using two focus groups to self report attitude and beliefs.
Existing COPD Clinical care operations within a variety of primary care practices. | Baseline to 2 years
  COPD clinical care operations at various practices will be assessed using two focus groups to self report current COPD clinical care operations within primary care clinicians own practices.
Existing COPD Clinical care operations within a variety of primary care practices. | Baseline to 2 years
  Details of COPD clinical care operations at various practices will be assessed using a questionnaire to self report current COPD clinical care operations within primary care clinicians own practices.
Primary care clinician attitudes and beliefs about screening and diagnostic assessment strategies of respiratory care and communication within their current practice. | Baseline to 2 years
  Primary care clinician attitudes and beliefs regarding screening and diagnostic assessment strategies and communication within their current practice will be assessed using two focus groups to self report attitude and beliefs.
Primary care clinician attitudes and beliefs about screening and diagnostic assessment strategies of respiratory care and communication within their current practice. | Baseline to 2 years
  Primary care clinician attitudes and beliefs regarding screening and diagnostic assessment strategies and communication within their current practice will be assessed using a prescriber questionnaire to self report attitude and beliefs.
Patient comprehension of CAPTURE tool instructions and questions. | Baseline to 2 years
  Patient comprehension of CAPTURE tool instructions and questions will be assessed using a CAPTURE opinion survey to self report comprehension.
Patient ease of completion of the CAPTURE tool. | Baseline to 2 years
  Patients' ease of completion of the CAPTURE tool will be assessed using a CAPTURE opinion survey to self report ease of completion.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - LANet, Los Angeles, California
  - High Plains Research Network, Aurora, Colorado
  - COPD Foundation, Miami, Florida
  - Atrium Healthcare, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Oregon Rural Practice-based Research Network (ORPRN), Portland, Oregon

IPD SHARING:
Plan to Share IPD: No